CLINICAL TRIAL: NCT03442582
Title: A Prospective Observational Safety Study on Pregnancy Outcomes in Women Immunized With Afluria, a Seasonal Influenza Vaccine, During Pregnancy
Brief Title: Afluria Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Other Study IDs: CSLCT-OBS-17-15
Record Dates: First submitted 2017-11-21; First posted 2018-02-22 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Influenza, Human; Pregnancy; Birth Defect
MeSH Terms: conditions — Influenza, Human; Congenital Abnormalities | interventions — Afluria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Afluria: Afluria exposure in pregnancy
  Interventions: Biological: Afluria Influenza Vaccine

INTERVENTIONS:
Biological: Afluria Influenza Vaccine — Afluria is a seasonal influenza vaccine
  Vaccine exposure in routine care (no vaccination per protocol)
  Other Names: Afluria

SUMMARY:
The study is a population based prospective cohort study designed to collect data on pregnancy outcomes and events of interest among women immunized with Afluria during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Enrollment and data collection will be coordinated through a coordination center (CC). The minimum eligibility criteria required for enrollment are as follows:

* Sufficient information to confirm that the exposure of interest occurred during pregnancy and at which date.
* Sufficient information to determine whether it concerns a prospectively enrolled subject, since retrospective cases are ineligible for enrollment.
* Reporter (e.g. HCP) contact information to allow for follow-up

Exclusion Criteria:

* N/A

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include pregnant women within the US who were immunized with Afluria as part of routine care at any time during pregnancy. Eligible pregnant women may self-enroll or voluntarily be enrolled by their HCP.
  Women under 18 can be included in the study as long as parental consent can be obtained, according to IRB requirements and local laws and regulations.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Safety Objective: Number of cases for pregnancy outcomes among women immunized as part of routine care with Afluria, a seasonal influenza vaccine, during pregnancy. | From time of enrollment during pregnancy to time of delivery or pregnancy termination; a follow-up period of up to 40 weeks
  Pregnancy outcomes will be reported as one of the following: live birth, stillbirth, spontaneous abortion and elective termination
Safety Objective: Number of cases with events of major congenital malformations among women immunized as part of routine care with Afluria, a seasonal influenza vaccine, during pregnancy. | From time of enrollment during pregnancy to time of delivery or pregnancy termination; a follow-up period of up to 40 weeks
Safety Objective: Number of cases of events of preterm birth among women immunized as part of routine care with Afluria, a seasonal influenza vaccine, during pregnancy. | From time of enrollment during pregnancy to time of delivery or pregnancy termination; a follow-up period of up to 40 weeks
Safety Objective: Number of cases of events of low birth weight among women immunized as part of routine care with Afluria, a seasonal influenza vaccine, during pregnancy. | From time of enrollment during pregnancy to time of delivery or pregnancy termination; a follow-up period of up to 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Head Epidemiology, Study Director — Seqirus
Locations (1):
- Syneos Health, Wilmington, North Carolina, United States